CLINICAL TRIAL: NCT06558409
Title: Safer Still (EP3)- An Interactive Intervention Adjunct to Traditional Care for Adolescents Who Are Discharged From Psychiatric Hospitals and Living in Households Where Firearms Are Stored Unsafely.
Brief Title: Safer Still (Exploratory Project 3)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jeff Bridge (Other)
Collaborators: Ohio Chapter American Academy of Pediatrics (Other)
Responsible Party: Sponsor-Investigator, Jeff Bridge, Principal Investigator: Jeffrey A Bridge, PhD,Abigail Wexner Research Institute at NCH, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00002773
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Suicide Prevention
Keywords: Firearms safety; Lethal means prevention; Safe storage of firearms and medication; Mobile application; Interactive intervention; Firearm storage behavior; Behavioral economics; Behavioral nudges; Lethal means restriction; Medication storage practices
MeSH Terms: conditions — Suicide Prevention | interventions — Economics, Behavioral

STUDY DESIGN:
Intervention Model Description: 80 families will be randomly assigned to either the Safer Still intervention (n=40) or EUC (n=40) in a parallel groups design. A stratified randomization procedure will balance the groups of participating parents on recruitment site.
Who Masked: Participant
Masking Description: Like the intervention Safer Still web-based program, the control website will be branded with a Nationwide Children's Hospital affiliation, as opposed to an outside organization that will be less familiar to the central Ohio sample. The control website will NOT feature these three behavioral economic strategies--namely (a) multiple suggested alternatives for means restriction, (b) requests to justify inaction regarding means restriction, and (c) normative feedback about means restriction.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Safer Still Intervention (Experimental): Investigators will present parents with suggested alternatives for restricting lethal means, particularly firearms and medications with high toxicity in overdose. Investigators will present multiple options for restricting access as opposed to just one alternative that may be deemed unreasonable by a family. Investigators will generate these options based upon the expertise of the study's lethal means consultant. Second, the mobile technology platform will provide weekly prompts about means restriction. Parents who have not restricted access to lethal means will be asked to document their reasons for inaction-a justification for not following safe storage practices. Third, the mobile technology platform will provide descriptive normative data regarding means restriction to those who have not secured these items
  Interventions: Behavioral: " Safer Still " Interactive Intervention
- Enhanced Usual Care (EUC) (Placebo Comparator): Families randomly assigned to the control condition will receive a psychological placebo that will feature an education only website developed by NCH's web design team. This website will cover warning signs for suicide, the leading methods of suicide - so that both conditions have content that features information about firearms - and locating professional help. Like the intervention Safer Still web-based program, the control website will be branded with a Nationwide Children's Hospital affiliation, as opposed to an outside organization that will be less familiar to the central Ohio sample. The control website will NOT feature these three behavioral economic strategies--namely (a) multiple suggested alternatives for means restriction, (b) requests to justify inaction regarding means restriction, and (c) normative feedback about means restriction.
  Interventions: Other: Enhanced Usual Care (EUC):

INTERVENTIONS:
Behavioral: " Safer Still " Interactive Intervention — An interactive intervention will be developed to help promote safe storage of firearms during the critical period immediately following high-risk care transitions.
  Other Names: Interactive intervention; Lethal means restriction; Safe storage; Firearm storage; Medication storage; Behavioral economics; Suicide prevention
  Arms: Safer Still Intervention
Other: Enhanced Usual Care (EUC): — Families randomly assigned to the control condition will receive a psychological placebo that will feature an education only website developed by NCH's web design team. This website will cover warning signs for suicide, the leading methods of suicide - so that both conditions have content that features information about firearms - and locating professional help. The control website will NOT feature these three behavioral economic strategies--namely (a) multiple suggested alternatives for means restriction, (b) requests to justify inaction regarding means restriction, and (c) normative feedback about means restriction.
  Arms: Enhanced Usual Care (EUC)

SUMMARY:
The long-term goal is to decrease suicide and suicidal behaviors in at-risk youth through preventative interventions. Investigators propose to develop an interactive intervention ("Safer Still") to help promote safe storage of firearms during the critical period immediately following high-risk care transitions. The objective of this study is to develop and test the Safer Still intervention as an efficient adjunct to traditional care for adolescents aged 12-17 years who are discharged from psychiatric hospitals and living in households where firearms are stored unsafely.

DETAILED DESCRIPTION:
The objective of this study is to develop and test the Safer Still intervention as an efficient adjunct to traditional care for adolescents aged 12-17 years who are discharged from psychiatric hospitals and living in households where firearms are stored unsafely. Exploratory aims of the study are as follows: (1) Evaluate parental motivation to change firearm storage behavior as a potential mediator of the three-month intervention effect. Investigators hypothesize that higher change scores in the "action" stage of the readiness to change model1 at one month will mediate the intervention effect at three months; (2) Identify whether the response to the Safer Still intervention varies by adolescent history of suicide attempt and parental primary reason for firearm ownership at one and three months; and (3) Ascertain common parental reasons for declining to safely store firearms.

ELIGIBILITY:
Inclusion Criteria:

* Parent or legal guardian of an adolescent aged 12 to 17 years at time of consent
* Have a child who is receiving psychiatric inpatient, crisis, or emergency treatment at Nationwide Children's Hospital
* Indicate that at least one firearm is located in or around the residence of the adolescent and is stored unlocked, loaded, or both unlocked and loaded.
* Only one parent per household is permitted to participate to avoid contamination across the two study conditions.

Exclusion Criteria:

* Inability to speak/read English
* Lack access to a digital device (smartphone, iPad, tablet computer, desktop, laptop PC).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Household Lethal Means Survey (HLMS) | Baseline, One month and Three months
  The Household Lethal Means Survey (HLMS) asks the parent to indicate whether there are any guns kept in or around the home, and if so to describe how the gun(s) and ammunition are stored. The HLMS will be supplemented with three questions from the 2018 California Safety and Well-Being Survey. These three questions address reasons for firearm ownership, loaded handgun carrying in the past 30 days, and high-capacity magazine ownership. At follow-up, the study survey assesses whether and how firearm ownership and storage practices changed since baseline. Similar questions at baseline and follow-up are asked about lethal medications.

SECONDARY OUTCOMES:
Stages of Change Questionnaire (SOCQ) | Baseline, One month, and Three months
  Readiness to change firearm and medication storage practices will be assessed using the Stages of Change Questionnaire (SOCQ), a psychometrically sound 12-item self-report measure ( 5-point Likert scale; -2 = "Strongly Disagree"; +2 = " Strongly Agree"). The scale will be used to measure the four stages of change (Pre-contemplation, Contemplation, Action, and Maintenance). Items numbered 1,3,6,10 Precontemplation, items numbered 2,4,7,11 = Contemplation and items numbered 5,8,9,12 = Action.
  A negative scale score reflects an overall disagreement with items measuring the stage of change, whereas a positive score represents overall agreement. The highest scale score represents the Stage of Change Designation.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Bridge, Ph.D., Principal Investigator — Nationwide Children's Hospital; Jack Stevens, Ph.D., Principal Investigator — Nationwide Children's Hospital
Locations (2):
- United States (2):
  - Nationwide Children's Hospital, Columbus, Ohio
  - Nationwide Children's Hospital Behavioral Health Pavillion, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, Analytic Code
Access Criteria: Researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal. Proposals should be directed tojeff.bridge@nationwidechildrens.org. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years after publication at a web address to be determined.

REFERENCES:
- [Background] Prochaska JO, Norcross JC. Stages of change. Psychotherapy. 2001;38(4):443-448
- [Background] Goldacre M, Seagroatt V, Hawton K. Suicide after discharge from psychiatric inpatient care. Lancet. 1993 Jul 31;342(8866):283-6. doi: 10.1016/0140-6736(93)91822-4. PMID 8101307
- [Background] Geddes JR, Juszczak E, O'Brien F, Kendrick S. Suicide in the 12 months after discharge from psychiatric inpatient care, Scotland 1968-92. J Epidemiol Community Health. 1997 Aug;51(4):430-4. doi: 10.1136/jech.51.4.430. PMID 9328552
- [Background] Chung DT, Ryan CJ, Hadzi-Pavlovic D, Singh SP, Stanton C, Large MM. Suicide Rates After Discharge From Psychiatric Facilities: A Systematic Review and Meta-analysis. JAMA Psychiatry. 2017 Jul 1;74(7):694-702. doi: 10.1001/jamapsychiatry.2017.1044. PMID 28564699
- [Background] Olfson M, Marcus SC, Bridge JA. Focusing suicide prevention on periods of high risk. JAMA. 2014 Mar 19;311(11):1107-8. doi: 10.1001/jama.2014.501. No abstract available. PMID 24515285
- [Background] Centers for Disease Control and Prevention. National Center for Injury Prevention and Control. Web-based Injury Statistics Query and Reporting System (WISQARS) [online]. [Last accessed, 5/9/20]. Source of data from WISQARS is the National Vital Statistics System from the National Center for Health Statistics. Available from URL: www.cdc.gov/ncipc/wisqars. Published 2018. Accessed.
- [Background] Office of the Surgeon General (US); National Action Alliance for Suicide Prevention (US). 2012 National Strategy for Suicide Prevention: Goals and Objectives for Action: A Report of the U.S. Surgeon General and of the National Action Alliance for Suicide Prevention. Washington (DC): US Department of Health & Human Services (US); 2012 Sep. Available from http://www.ncbi.nlm.nih.gov/books/NBK109917/ PMID 23136686
- [Background] Meeker D, Linder JA, Fox CR, Friedberg MW, Persell SD, Goldstein NJ, Knight TK, Hay JW, Doctor JN. Effect of Behavioral Interventions on Inappropriate Antibiotic Prescribing Among Primary Care Practices: A Randomized Clinical Trial. JAMA. 2016 Feb 9;315(6):562-70. doi: 10.1001/jama.2016.0275. PMID 26864410
- [Background] Wang SY, Groene O. The effectiveness of behavioral economics-informed interventions on physician behavioral change: A systematic literature review. PLoS One. 2020 Jun 4;15(6):e0234149. doi: 10.1371/journal.pone.0234149. eCollection 2020. PMID 32497082
- [Background] Bauer BW, Capron DW. How Behavioral Economics and Nudges Could Help Diminish Irrationality in Suicide-Related Decisions. Perspect Psychol Sci. 2020 Jan;15(1):44-61. doi: 10.1177/1745691619866463. Epub 2019 Nov 7. PMID 31697611
- [Background] Davis M, Wolk CB, Jager-Hyman S, Beidas RS, Young JF, Mautone JA, Buttenheim AM, Mandell DS, Volpp KG, Wislocki K, Futterer A, Marx D, Dieckmeyer EL, Becker-Haimes EM. Implementing nudges for suicide prevention in real-world environments: project INSPIRE study protocol. Pilot Feasibility Stud. 2020 Sep 26;6:143. doi: 10.1186/s40814-020-00686-y. eCollection 2020. PMID 32995040
- [Background] Horowitz LM, Wharff EA, Mournet AM, Ross AM, McBee-Strayer S, He JP, Lanzillo EC, White E, Bergdoll E, Powell DS, Solages M, Merikangas KR, Pao M, Bridge JA. Validation and Feasibility of the ASQ Among Pediatric Medical and Surgical Inpatients. Hosp Pediatr. 2020 Sep;10(9):750-757. doi: 10.1542/hpeds.2020-0087. PMID 32826283
- [Background] Stiffman AR, Horwitz SM, Hoagwood K, Compton W 3rd, Cottler L, Bean DL, Narrow WE, Weisz JR. The Service Assessment for Children and Adolescents (SACA): adult and child reports. J Am Acad Child Adolesc Psychiatry. 2000 Aug;39(8):1032-9. doi: 10.1097/00004583-200008000-00019. PMID 10939232
- [Background] Horwitz SM, Hoagwood K, Stiffman AR, Summerfeld T, Weisz JR, Costello EJ, Rost K, Bean DL, Cottler L, Leaf PJ, Roper M, Norquist G. Reliability of the services assessment for children and adolescents. Psychiatr Serv. 2001 Aug;52(8):1088-94. doi: 10.1176/appi.ps.52.8.1088. PMID 11474056
- [Background] Bellis JM. The transtheoretical model of change applied to psychotherapy: A psychometric assessment of related instruments.: Dissertation Abstracts International, 54B, 3846. (UMI No. AAC9332421); 1994.
- [Background] Lewis CC, Simons AD, Silva SG, Rohde P, Small DM, Murakami JL, High RR, March JS. The role of readiness to change in response to treatment of adolescent depression. J Consult Clin Psychol. 2009 Jun;77(3):422-8. doi: 10.1037/a0014154. PMID 19485584
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Achenbach TM, Dumenci L, Rescorla LA. DSM-oriented and empirically based approaches to constructing scales from the same item pools. J Clin Child Adolesc Psychol. 2003 Sep;32(3):328-40. doi: 10.1207/S15374424JCCP3203_02. PMID 12881022
- [Background] Richardson LP, McCauley E, Grossman DC, McCarty CA, Richards J, Russo JE, Rockhill C, Katon W. Evaluation of the Patient Health Questionnaire-9 Item for detecting major depression among adolescents. Pediatrics. 2010 Dec;126(6):1117-23. doi: 10.1542/peds.2010-0852. Epub 2010 Nov 1. PMID 21041282
- [Background] Nguyen TD, Attkisson CC, Stegner BL. Assessment of patient satisfaction: development and refinement of a service evaluation questionnaire. Eval Program Plann. 1983;6(3-4):299-313. doi: 10.1016/0149-7189(83)90010-1. PMID 10267258
- [Background] Posner K, Brent D, Lucas C, et al. Columbia-Suicide Severity Rating Scale (C-SSRS) New York State Psychiatric Institute https://cssrs.columbia.edu/wp-content/uploads/C-SSRS_Pediatric-SLC_11.14.16.pdf
- [Background] Pierce DW. Suicidal intent in self-injury. Br J Psychiatry. 1977 Apr;130:377-85. doi: 10.1192/bjp.130.4.377. PMID 870128
- [Background] Association AP. DSM-5-TR Online Assessment Measures. Accessed July 21, 2022. https://www.psychiatry.org/psychiatrists/practice/dsm/educational-resources/assessment-measures
- See also: PhenX Toolkit: Mental Health Research Core Tier 1 Demographic and Social Environment Measures — https://www.phenxtoolkit.org/sub-collections/view/1
- See also: PhenX Toolkit: Suicide Specialty Collection - Access to Lethal Means Measure — https://www.phenxtoolkit.org/toolkit/?add[]=641001